CLINICAL TRIAL: NCT04686526
Title: Development of a Wearable Electrocardiogram Monitoring Device and Smartphone Application in Perioperative Pain Management
Brief Title: Wearable Electrocardiogram Monitoring Device and Smartphone Application in Perioperative Pain Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-2489
Record Dates: First submitted 2020-10-26; First posted 2020-12-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
Keywords: heart rate variability; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a wearable electrocardiograph monitoring device and smartphone application in perioperative pain management, also to evaluate relationship between postoperative pain and heart rate variability.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study implementing wearable electrocardiogram (ECG) monitor device and smartphone application in perioperative pain management. Patients undergoing major abdominal surgical procedures will be recruited to wear a ECG monitor device from the day before surgery until 1-3days after surgery. Patients will report their condition of pain twice daily on the corresponding smartphone application based on a structured and visualized pain report module. Patients will receive a telephone follow-up 30/60/90/365 days after surgery for assessment of postoperative chronic pain. A pilot study will be conducted to evaluate acceptability, safety and feasibility of the device and application using system usability scale and comprehensive product quality assessment. Further study will be conducted to evaluate the relationship between postoperative acute and chronic pain and heart rate variability (HRV) acquired from ECG device.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing major abdominal surgical procedures;
* 18-65 years old;
* ASA classification: I-IV
* able to read and understand how to use the App after instruction；
* written informed consent obtained.

Exclusion Criteria:

* current participation in other mobile device research or perioperative pain research;
* inability to use the device;
* inability to obtain consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgical procedures in Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate to severe acute post-operative pain | Postoperative Day 1 to 3
  Visual Analogue Scale (VAS) value of patients will be assessed after surgery for three consecutive days, any VAS value ≥ 4 will be considered as an event of moderate to severe acute post-operative pain

SECONDARY OUTCOMES:
Incidence of chronic post-surgical pain | 1 year after surgery
  Patient's chronic pain condition will be assessed by Defense & Veterans Pain Rating Scale (DVPRS) score one year after surgery, a DVPRS score ≥5 is considered as an existence of chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Li Xu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China